CLINICAL TRIAL: NCT05098574
Title: A Pilot, Randomized, Placebo-Controlled Trial Evaluating the Treatment of Premenstrual Dysphoric Disorder with Oral Contraceptives in Bipolar Disorder.
Brief Title: Oral Contraceptives for Treating Premenstrual Dysphoric Disorder in Bipolar Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Hamilton Academic Health Sciences Organization (Other); McMaster University (Other)
Responsible Party: Principal Investigator, Benicio Frey, Psychiatrist/ Professor, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BDPMDD01
Record Dates: First submitted 2021-07-14; First posted 2021-10-28 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Premenstrual Dysphoric Disorder; Bipolar Disorder
Keywords: bipolar disorder; premenstrual dysphoric disorder
MeSH Terms: conditions — Premenstrual Dysphoric Disorder; Bipolar Disorder | interventions — drospirenone and ethinyl estradiol combination; drospirenone; Ethinyl Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined oral contraceptive (3mg drospirenone/ 0.02mg ethinyl estradiol) (Experimental): Continuous treatment with 3mg drospirenone/ 0.02mg ethinyl estradiol for 12 weeks
  Interventions: Drug: Yaz
- Placebo (Placebo Comparator): Continuous treatment with placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Yaz — Continuous treatment with 3mg drospirenone/ 0.02mg ethinyl estradiol for 12 weeks
  Other Names: 3mg drospirenone/ 0.02mg ethinyl estradiol
  Arms: Combined oral contraceptive (3mg drospirenone/ 0.02mg ethinyl estradiol)
Drug: Placebo — Appearance, packaging, and labeling of placebo will be matched to their active counterpart.
  Arms: Placebo

SUMMARY:
This study is a pilot, randomized, placebo-controlled trial evaluating the treatment of Premenstrual Dysphoric Disorder comorbid with Bipolar Disorder using combined oral contraceptives.

Lay Summary:

This study is being done with the hope of finding a safe and effective treatment for individuals who experience both bipolar disorder and severe premenstrual symptoms. As part of this clinical trial, participants will receive either a combined oral contraceptive (i.e. oral birth control pills) as a treatment for severe premenstrual symptoms or a placebo (a pill without any active components - similar to a sugar pill). People that are enrolled in this study will either receive the treatment or the placebo for a period of 90 days. During this time, people that are participating in the study will fill out some questionnaires, and their mental and physical health will be monitored by the study physicians.

One of the goals of this study is to also understand whether it is feasible (practical) to do a larger clinical trial using this treatment in this group of people.

ELIGIBILITY:
Inclusion Criteria:

* 16-45 years of age
* Diagnosis of BD (clinically euthymic) according to the DSM-5
* Diagnosis of PMDD according to the DSM-5
* Regular menstrual cycles
* No contraindication to use oral contraceptives
* Capable of consent for treatment

Exclusion Criteria:

* Smoking and over the age of 35
* Current or recent (last month) use of systemic estrogen or progesterone treatment
* Severe reactions to hormone treatment
* Pregnant or breastfeeding
* Current substance use disorder
* Oophorectomy or hysterectomy
* Current unstable medical conditions
* History of current or past breast cancer, pancreatitis, migraines or blood clotting disorders.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Feasibility outcome: treatment compliance | 12 weeks
  Treatment compliance - assessed via number and percentage of treatment pills taken
Feasibility outcome: retention rates | 12 weeks
  Retention rates - number and percentage of people who remain in the study once randomized
Feasibility outcome: recruitment rate (monthly) | 2 years
  Recruitment rate (monthly) - number of participants per month
Feasibility outcome: recruitment capacity | 2 years
  Recruitment capacity - total number of participants randomized and enrolled
Feasibility outcome: screening rates (monthly) | 2 years
  Screening rates (monthly) - number screened; number enrolled as a percentage of number screened
Feasibility outcome: duration of assessment process | Screening
  Duration of assessment process - mean in hours from start to finish for each visit
Feasibility outcome: duration of assessment process | Baseline
  Duration of assessment process - mean in hours from start to finish for each visit
Feasibility outcome: duration of assessment process | Week 4
  Duration of assessment process - mean in hours from start to finish for each visit
Feasibility outcome: duration of assessment process | Week 8
  Duration of assessment process - mean in hours from start to finish for each visit
Feasibility outcome: duration of assessment process | Week 12
  Duration of assessment process - mean in hours from start to finish for each visit
Feasibility outcome: safety of use of oral contraceptives in this population | Week 4
  Safety of use of oral contraceptives in this population - adverse events reported, onset of mood episodes (assessed by clinicians)
Feasibility outcome: safety of use of oral contraceptives in this population | Week 8
  Safety of use of oral contraceptives in this population - adverse events reported, onset of mood episodes (assessed by clinicians)
Feasibility outcome: safety of use of oral contraceptives in this population | Week 12
  Safety of use of oral contraceptives in this population - adverse events reported, onset of mood episodes (assessed by clinicians)
Feasibility outcome: tolerability | Week 4
  Tolerability - assessed as percentage dropped out after randomization due to adverse events
Feasibility outcome: tolerability | Week 8
  Tolerability - assessed as percentage dropped out after randomization due to adverse events
Feasibility outcome: tolerability | Week 12
  Tolerability - assessed as percentage dropped out after randomization due to adverse events
Feasibility outcome: response rates | Week 12
  Response rates - response will be defined as 50% decrease from baseline symptom change from late luteal to follicular phase; remission will be defined as number and percentage of responders who no longer need DSM-5 criteria for PMDD
Feasibility outcome: estimated treatment effect | Week 12
  Estimated treatment effect - mean percent change from baseline to post-treatment in percent change on the MAC-PMSS from late luteal to follicular phase
Feasibility outcome: variance of the treatment effect | Week 12
  Variance of the treatment effect - standard deviation of above measure.

CONTACTS AND LOCATIONS:
Overall Officials: Benicio N Frey, MD, MSc,PhD, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma S, Song SJ. Oral contraceptives containing drospirenone for premenstrual syndrome. Cochrane Database Syst Rev. 2023 Jun 23;6(6):CD006586. doi: 10.1002/14651858.CD006586.pub5. PMID 37365881